CLINICAL TRIAL: NCT02146989
Title: Upper Extremity Strength in Children and Adolescents With and Without Unilateral Cerebral Palsy
Brief Title: Upper Extremity Strength in Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Maastricht University (Other); Adelante, Centre of Expertise in Rehabilitation and Audiology (Other); Revant (Unknown); Tolbrug (Unknown); Libra Zorggroep (Unknown); VieCuri Medical Centre (Other)
Responsible Party: Sponsor
Other Study IDs: NL45430.068.13
Record Dates: First submitted 2014-05-21; First posted 2014-05-26 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; child; upper extremity; strength, reproducibility
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cerebral Palsy: Children and adolescents with spastic unilateral Cerebral Palsy (with perinatal acquired hypoxic ischemic incidents), aged 7 to 18 years, MACS levels I-III.
  Interventions: Other: reproducibility of upper extremity strength measurements
- Healthy controls: Children and adolescents without Cerebral Palsy
  Interventions: Other: reproducibility of upper extremity strength measurements

INTERVENTIONS:
Other: reproducibility of upper extremity strength measurements — inter-rater reliability and test-retest reliability
  Other Names: Hand Held Dynamometry; E-link system; functional strength measurements

SUMMARY:
Rationale:

Children with Cerebral Palsy (CP) experience limitations in motor activities and participation in the community, predominantly caused by impairments in muscle function. Aside from abnormal posturing due to spasticity, muscle weakness can significantly contribute to impaired muscle function and there is increasing evidence that muscle weakness significantly impairs upper limb motor function and ability to perform manual tasks in children with CP. Studies in the last decade have shown that muscle weakness, not spasticity, is the greatest limiting factor of motor function in children with CP. Furthermore, there is increasing evidence that the strength in the upper extremities of children with CP is less compared to their typically developing peers (TDP). A systematic review focused on the psychometric properties of strength measurement instruments has shown that the number of studies investigating psychometric properties of strength measurement instruments is limited and that the methodological quality of these studies is low.

Aim:

The present study aims to investigate the reproducibility of the following three isometric strength measurements in the upper extremity of children and adolescents with unilateral CP as well as in TDP: Hand Held Dynamometry (HHD), pinch and grip strength using the E-link system and functional strength. To study to which extent upper extremity strength, both in the affected side and the non-affected side, differs from the strength in the upper extremities of TDP, these measurements will also be performed by children without neurological problems.

Study Design:

A cross-sectional study in which the reproducibility of three strength measurement instruments, i.e. HHD, E-link and Functional strength, will be investigated in children and adolescents with unilateral CP and TDP.

Population:

Children with unilateral spastic CP (with perinatal acquired hypoxic ischemic incidents), aged 7 to 18 years, Manual Ability Classification System (MACS) levels I-III, who are mentally able to perform the measurements will be included and TDP.

Outcome measures:

The most important psychometric property in strength measurement instruments is reproducibility. Reproducibility will be investigated using the following factors: Intraclass Correlation Coefficient (ICC), Limits of Agreement (LOA), Standard Error of Measurement (SEM) and the Smallest Detectable Difference (SDD). Reference values will be determined using the Generalised Additive Models for Location, Scale, and Shape (GAMLSS) method.

ELIGIBILITY:
Inclusion Criteria CP:

* Children with unilateral spastic CP (with perinatal acquired hypoxic ischemic incidents),
* aged 7 to 18 years,
* MACS levels I-III,
* mentally able to perform the measurements

Inclusion criteria Healthy Controls:

* children attending primary or secondary school
* agd 7 to 18 years

Exclusion Criteria CP:

* Surgical intervention <6 months
* Botulinum Toxin A treatment in the upper extremity < 6 months
* contractures in the upper extremity that might interfere with task performance

Exclusion criteria Healthy Controls:

* muscle disease
* lesion, fracture or cast < 6 months

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Spastic unilateral Cerebral Palsy and Healthy Controls
Sampling Method: Non-Probability Sample
Enrollment: 370 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2018-03-19 (Actual); Study Completion 2018-03-19 (Actual)

PRIMARY OUTCOMES:
Inter-rater and test-retest reliability of HHD expressed as ICC value | t1 (base-line) and t1 (2-3 weeks later)
  The intraclass correlation coefficient (ICC) is commonly used in the assessment of consistency or reproducibility of quantitative measurements made by different observers measuring the same quantity.
Inter-rater and test-retest reliability of E-link expressed as ICC value | t1 (base-line) and t1 (2-3 weeks later)
  The intraclass correlation coefficient (ICC) is commonly used in the assessment of consistency or reproducibility of quantitative measurements made by different observers measuring the same quantity.
Inter-rater and test-retest reliability of functional strength measurements expressed as ICC value | t1 (base-line) and t1 (2-3 weeks later)
  The intraclass correlation coefficient (ICC) is commonly used in the assessment of consistency or reproducibility of quantitative measurements made by different observers measuring the same quantity.
Inter-rater and test-retest agreement of HHD expressed as Limits of Agreement | t1 (base-line) and t1 (2-3 weeks later)
  The limits of agreement (LOA) provide insight into how much random variation may be influencing the ratings. If the raters tend to agree, the differences between the raters' observations will be near zero. If one rater is usually higher or lower than the other by a consistent amount, the bias (mean of differences) will be different from zero. If the raters tend to disagree, but without a consistent pattern of one rating higher than the other, the mean will be near zero. Confidence limits (usually 95%) can be calculated for both the bias and each of the limits of agreement.
Inter-rater and test-retest agreement of E-Link expressed as Limits of Agreement | t1 (base-line) and t1 (2-3 weeks later)
  The limits of agreement (LOA) provide insight into how much random variation may be influencing the ratings. If the raters tend to agree, the differences between the raters' observations will be near zero. If one rater is usually higher or lower than the other by a consistent amount, the bias (mean of differences) will be different from zero. If the raters tend to disagree, but without a consistent pattern of one rating higher than the other, the mean will be near zero. Confidence limits (usually 95%) can be calculated for both the bias and each of the limits of agreement.
Inter-rater and test-retest agreement of functional measurements expressed as Limits of Agreement | t1 (base-line) and t1 (2-3 weeks later)
  The limits of agreement (LOA) provide insight into how much random variation may be influencing the ratings. If the raters tend to agree, the differences between the raters' observations will be near zero. If one rater is usually higher or lower than the other by a consistent amount, the bias (mean of differences) will be different from zero. If the raters tend to disagree, but without a consistent pattern of one rating higher than the other, the mean will be near zero. Confidence limits (usually 95%) can be calculated for both the bias and each of the limits of agreement.

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne JM Janssen-Potten, PhD, Principal Investigator — Adelante, Centre of Expertise in Rehabilitation and Audiology
Locations (9):
- Netherlands (9):
  - Adelante, Hoensbroek, Limburg
  - Tolbrug, 's-Hertogenbosch
  - Klimmendaal, Arnhem
  - Revant, Breda
  - Libra Zorggroep, Eindhoven
  - Rijnlands Revalidatie Centrum, Leiden
  - St. Maartenskliniek, Nijmegen
  - Sophie Revalidatie, The Hague
  - Viecuri Medical Centre, Venlo